CLINICAL TRIAL: NCT04241718
Title: A Feasibility Study on Ultrafiltration and Blood Volume Measurements
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Nuwellis, Inc. (Industry)
Collaborators: Daxor Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLIN06477
Record Dates: First submitted 2019-11-25; First posted 2020-01-27 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Acute Decompensated Heart Failure; Fluid Overload
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single-arm (Other): No comparator, placebo, or randomization
  Interventions: Device: Aquadex FlexFlow System and BVA-100

INTERVENTIONS:
Device: Aquadex FlexFlow System and BVA-100 — Aquapheresis therapy with Aquadex FlexFlow System and Blood Volume Measurement with BVA-100

SUMMARY:
The objective of this feasibility study is to characterize the performance of the Aquadex FlexFlow® System with the hematocrit (HCT) feature in conjunction with Daxor's blood volume analyzer (BVA-100). The study will monitor blood volume changes during ultrafiltration (UF) therapy as a potential means to guide the removal of fluid in subjects hospitalized with acute decompensated heart failure (ADHF).

DETAILED DESCRIPTION:
The study will measure blood volumes at various time intervals using the BVA-100 for comparison to corresponding readings of hematocrit (HCT) levels from the Aquadex FlexFlow HCT sensor. Establishing a correlation between BVA measurements (off-line measurements) and HCT sensor measurements (on-line measurements) may enable the use of the BVA-100 to guide ultrafiltration therapy by the Aquadex system for fluid removal.

BVA-100 measurements would be used at baseline to accurately determine patient suitability for fluid removal and while HCT measurements would be used to monitor blood volume changes during ultrafiltration therapy, potentially guiding the removal of fluid in subjects hospitalized with ADHF.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Subject or legally authorized representative is able to provide appropriate consent to participate
3. Hospitalized for ADHF with fluid overload as indicated by at least two of the following:

   1. Pitting edema ≥ 2+ of the lower extremities
   2. Jugular venous distention > 8 cm
   3. Pulmonary edema/pleural effusion on chest x-ray
   4. Paroxysmal nocturnal dyspnea or ≥ two- pillow orthopnea
   5. Respiration rate ≥ 20 per minute

Exclusion Criteria:

1. Unable or unwillingness to provide informed consent or to comply with study requirements
2. Subject who is pregnant
3. Acute coronary syndrome
4. Known bilateral renal artery stenosis
5. Serum creatinine > 3.0 mg/dL at the time of presentation
6. Subject receiving ongoing active treatment with diuretics (up to 2 doses of IV diuretics are permitted before initiation of ultrafiltration therapy)
7. Systolic blood pressure ≤ 90 mmHg
8. Poor or unattainable central access
9. Has bleeding disorder
10. Contraindications to systemic anticoagulation
11. Allergic to iodine, albumin, or iodinated I-131 albumin
12. Active myocarditis or hypertrophic obstructive cardiomyopathy
13. Severe uncorrected valvular stenosis
14. Complex congenital heart disease
15. Systemic infection
16. Previous organ transplant
17. Enrollment in other clinical trials
18. Life expectancy ≤ 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
1. Evaluate changes in blood volume as measured by BVA from before initiation until completion of extracorporeal fluid removal by ultrafiltration | Through study procedure completion, average of 2 weeks
  BVA will be used to evaluate changes in blood volume from baseline (i.e., before initiation) until completion of extracorporeal fluid removal by ultrafiltration.
2. Evaluate if changes in blood volume, as measured by BVA, correlate with changes in HCT as measured by the device embedded in the Aquadex FlexFlow System ultrafiltration device | Through study procedure completion, average of 2 weeks
  A correlation between BVA measured change in blood volume to changes in hematocrit (HCT) as measured by the online HCT sensor embedded in the Aquadex Flexflow system will be determined.
3. Evaluate the temporal relationship between changes in blood volume, as measured by BVA , and changes in clinical signs and symptoms of fluid overload | Through study procedure completion, average of 2 weeks
  Temporal relationship between blood volume change (as measured by the BVA) and changes in clinical signs and symptoms of fluid overload will be evaluated.
4. Evaluate the temporal relationship between changes in HCT, as measured by Aquadex HCT, and changes in clinical signs and symptoms of fluid overload | Through study procedure completion, average of 2 weeks
  Temporal relationship between HCT change (as measured by Aquadex HCT sensor) and changes in clinical signs and symptoms of fluid overload will be evaluated.
5. Total net fluid loss prior to hospital discharge | Daily during study procedure, average of 2 weeks
  The total net fluid removed during the ultrafiltration therapy will be evaluated.
6. Change in urinary sodium concentration from baseline to ultrafiltration completion | Through study procedure completion, average of 2 weeks
  Urinary sodium concentration profile from baseline to ultrafiltration completion will be evaluated.
7. Change in biomarkers from baseline until discharge: | through study completion, average of 2 weeks
  * Comprehensive Metabolic Panel (CMP)/Basic Metabolic Panel (BMP)
  * N-terminal proB- type natriuretic peptide (NT-proBNP)
  * Troponin-I
  * Urine Nephrocheck
8. Adverse events of special interest | through study completion, average of 1 year
  * Acute coronary syndrome
  * Bleeding (requiring blood transfusion or drop of hemoglobin >3g/dl)
  * Catheter-related bloodstream infections
  * Hypotension necessitating intervention

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosa Costanzo, MD, Principal Investigator — Edward Hospital Center for Advanced Heart Failure; Maria Rosa Costanzo, MD, Principal Investigator — Edward-Elmhurst Health System
Locations (1):
- Midwest Cardiovascular Institute, Naperville, Illinois, United States

IPD SHARING:
Plan to Share IPD: No